CLINICAL TRIAL: NCT02680379
Title: A Pilot Study Exploring the Safety and Synergistic Effect of a Minocycline/Lovastatin Combined Treatment on the Behavior of Individuals With Fragile X Syndrome; Validation of New Biochemical and Neurophysiological Markers (LovaMiX)
Brief Title: Combined Treatment of Minocycline and Lovastatin to Treat Individuals With Fragile X Syndrome
Acronym: LovaMiX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: FRAXA Research Foundation (Other)
Responsible Party: Principal Investigator, Francois Corbin, Dr Francois Corbin, MD, PHD, FRCPC, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-1177
Record Dates: First submitted 2016-01-25; First posted 2016-02-11 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Fragile X Syndrome
Keywords: Fragile X Syndrome; Autism; FMR1; FRAXA
MeSH Terms: conditions — Fragile X Syndrome; Autistic Disorder | interventions — Minocycline; Lovastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Minocycline, then Minocycline/Lovastatin (Experimental): Participants will take minocycline then a combined treatment of minocycline/lovastatin for 3 months.
  Interventions: Drug: Minocycline, then Minocycline/Lovastatin
- Lovastatin, then Minocycline/Lovastatin (Experimental): Participants will lovastatin then a combined treatment of minocycline/lovastatin for 3 months
  Interventions: Drug: Lovastatin, then Minocycline/Lovastatin

INTERVENTIONS:
Drug: Minocycline, then Minocycline/Lovastatin — Participants of this group will take 1 tablet of minocycline 50mg daily for 4 weeks, minocycline 100mg for the following 4 weeks and finally a combined treatment of minocycline 100 mg and lovastatin 40mg for the following 12 weeks.
  Other Names: Minocin
  Arms: Minocycline, then Minocycline/Lovastatin
Drug: Lovastatin, then Minocycline/Lovastatin — Participants of this group will take 1 tablet of lovastatin 20 mg daily for 4 weeks, lovastatin 40 mg for the following 4 weeks and finally a combined treatment of minocycline 100 mg and lovastatin 40 mg for the following 12 weeks.
  Other Names: Mevacor
  Arms: Lovastatin, then Minocycline/Lovastatin

SUMMARY:
The purpose of this study is to determine whether Lovastatin, Minocycline and the combination Lovastatin/Minocycline are effective in treating behavioral symptoms in Fragile X individuals.

ELIGIBILITY:
Inclusion Criteria:

* Molecular diagnosis of fragile X syndrome
* The participant must be accompanied his parent, legal tutor or legal representative.
* Identify a caregiver who spends at least six hours per day with the participant (may be the parent, legal tutor, legal representative or an other person).
* IQ < 70
* ABC-C score > 20
* CGI-Severity score ≥ 4

Exclusion Criteria:

* Pregnant or breastfeeding participants
* Previous intolerance/allergy to statins, minocycline or tetracyclines
* Participants who have taken lovastatin or minocycline in the last 12 weeks
* Personal history of myopathy, myalgia or high creatine kinase (CK) levels
* Renal disease / liver disease / disturbed hepatorenal tests
* Participants taking more than three psychoactive medications (except anticonvulsants)
* Untreated or uncontrolled hypothyroidism
* Any other active medical condition
* Modification of psychoactive treatment in the last 6 weeks prior to randomization
* Participants under the age of 13 years who have incomplete formation of the crown of their teeth (except possibly their 3rd molars) as shown by panorex
* Concomitant use of prohibited drugs

  * Prohibited drugs include other hypolipemic including gemfibrozil (or other fibrates) and niacin (nicotinic acid), angiotensin converting enzyme (ACE), cyclosporine, danazol, amiodarone, verapamil and inhibitors P450 (CYP3A4) (itraconazole, ketoconazole, erythromycin, clarithromycin, telithromycin, inhibitors of HIV protease and nefazodone).

Ages: 8 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline Aberrant Behavior Checklist-Community (ABC-C) total score at 8,12 and 20 weeks | baseline, 8 weeks, 12 weeks, 20 weeks

SECONDARY OUTCOMES:
Clinical Global Impression Scale improvement (CGI-I) | baseline, 8 weeks, 12 weeks, 20 weeks
Change from baseline Social Responsiveness Scale (SRS) at 8 and 20 weeks | baseline, 8 weeks, 20 weeks
Anxiety, depression and mood scale (ADAMS), change from baseline to 8 and 20 weeks | baseline, 8 weeks, 20 weeks
Behavior Rating Inventory of Executive Function (BRIEF) | Before treatment and at the end of treatment (weeks 20)
Change from baseline Vineland II; adaptive behaviour scale at 20 weeks | baseline, 20 weeks

OTHER OUTCOMES:
(optional) Change in brain activity using Functional Magnetic Resonance Imaging (fMRI) at 8 and 20 weeks | baseline, 8 weeks, 20 weeks
  fMRI is a non-invasive method of assessing brain activity by detecting signal changes in blood flow and oxygenation known as BOLD (Blood-Oxygen-Level Dependent) contrast imaging.
(optional) Change in neurochemistry using Transcranial Magnetic Stimulation (TMS) at 8 and 20 weeks | baseline, 8 weeks, 20 weeks
  Using an unpainful magnetic stimulation on the primary motor cortex, TMS will be used to assess intracortical facilitation and inhibition, corresponding respectively to glutamate and GABAergic processes.

CONTACTS AND LOCATIONS:
Overall Officials: François Corbin, MD/PhD, Principal Investigator — Fragile X Clinic, Centre de recherche du CHUS
Locations (1):
- Centre de Recherche du CHUS, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Morin-Parent F, Champigny C, Cote S, Mohamad T, Hasani SA, Caku A, Corbin F, Lepage JF. Neurophysiological effects of a combined treatment of lovastatin and minocycline in patients with fragile X syndrome: Ancillary results of the LOVAMIX randomized clinical trial. Autism Res. 2024 Sep;17(9):1944-1956. doi: 10.1002/aur.3222. Epub 2024 Sep 9. PMID 39248107
- See also: Investigator profile — http://cr.chus.qc.ca/en/axes/mother-child/chercheurs/francois-corbin-m-d-ph-d/